CLINICAL TRIAL: NCT03089008
Title: Eccentric Exercise in Treatment of Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (KF) 01-157/98, (KF) 01-109/99; 1999-DP-65-RKF-11 [CTU]
Record Dates: First submitted 2016-08-25; First posted 2017-03-24 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Achillodynia
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eccentric exercises (Experimental): The patients were instructed to stand with straight legs on a small step, lift up on the toes, hereafter put the weight on the injured leg and slowly lower the heel as far as possible until they felt a maximal stretch of the calf muscles and/or the Achilles tendon. The exercises were repeated 15 times. Then the patients were told to repeat the exercises with semi-flexed knee. If possible the series should be repeated twice increasing to three times at each session. If pain decreased they should increase the load on the Achilles tendons by wearing a rug sack and increasing the weight of the rug sack by adding weights (5kg each). The patients were told that some pain was to be expected from the tendon during exercise, but that increasing daily pain or morning stiffness indicated that the exercises had been progressed too fast.
  Interventions: Other: Eccentric exercises
- Control treatment, stretching exercises (Other): The patients were instructed in standing stretching exercises of the gastrocnemius (straight leg) and soleus (bended knee). The stretch was slowly increased and maintained for 30s. This stretch was to be repeated five times during each session. The patients were instructed that the stretching should be pain free, although a small degree of unpleasantness was allowed.
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Other: Eccentric exercises
  Arms: Eccentric exercises
Other: Stretching exercises
  Arms: Control treatment, stretching exercises

SUMMARY:
The purpose of the present study is to examine the long-term effect of eccentric exercises compared with stretching exercises on patients with achillodynia.

DETAILED DESCRIPTION:
Patients with achillodynia for at least 3 months are randomly allocated to one of two exercise regimens. Exercise is performed daily for a 3-month period. Symptom severity is evaluated by tendon tenderness, ultrasonography, a questionnaire on pain and other symptoms, and a global assessment of improvement. Follow-up is performed at time points 3, 6, 9, 12 weeks and 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Pain in the Achilles tendon area with one of the two following findings. a) Distinct tenderness of Achilles tendon with no pain in the neighboring structures. b) Ultrasonographic changes defined as local thickening of the symptomatic tendon or a globally more than 2mm thicker tendon on the sick side.
2. Diffuse pain in the posterior region of the ankle with local tenderness of the Achilles tendon and ultrasonographic changes (as described above).

Exclusion Criteria:

1. Treatment of achillodynia with stretching or eccentric training for more than 2 weeks within the last 2 years.
2. Other injuries in the lower extremity or the knee, which by the examining doctor was evaluated to influence the evaluation of symptoms or the ability to perform the training program.
3. Acute symptoms with ultrasonographic changes consistent with a partial rupture of the tendon.
4. Age less than 18 years or over 70 years.
5. Previous operation on the tendon or steroid injections.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1999-01; Primary Completion 2000-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Manually assessed tenderness at inclusion | At inclusion
  The tenderness of the symptomatic tendons was determined manually by applying a moderate amount of pressure (about 1 kg) with the first and second finger on each side of the tendon. The tendon was palpated 0, 1, 3, 5, 7 and 10 cm proximal to the calcaneal insertion, and at each level the tenderness score was noted according to the subjects' answers of the pain perceived (0 = none, 1 = mild, 2 = moderate and 3 = severe).
Change in manually assessed tenderness after 12 weeks | 12 weeks
  The tenderness of the symptomatic tendons was determined manually by applying a moderate amount of pressure (about 1 kg) with the first and second finger on each side of the tendon. The tendon was palpated 0, 1, 3, 5, 7 and 10 cm proximal to the calcaneal insertion, and at each level the tenderness score was noted according to the subjects' answers of the pain perceived (0 = none, 1 = mild, 2 = moderate and 3 = severe).
Change in manually assessed tenderness after 39 weeks | 39 weeks
  The tenderness of the symptomatic tendons was determined manually by applying a moderate amount of pressure (about 1 kg) with the first and second finger on each side of the tendon. The tendon was palpated 0, 1, 3, 5, 7 and 10 cm proximal to the calcaneal insertion, and at each level the tenderness score was noted according to the subjects' answers of the pain perceived (0 = none, 1 = mild, 2 = moderate and 3 = severe).

CONTACTS AND LOCATIONS:
Overall Officials: Per Jessen, Study Chair
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan to share data.